CLINICAL TRIAL: NCT04444284
Title: A Randomized, Single-Blind, Placebo-Controlled, Dose-Escalation Phase 1b Study to Evaluate the Safety and Immunogenicity of an Intranasal Live Attenuated Respiratory Syncytial Virus (RSV) Vaccine in Seropositive Young Children
Brief Title: Study of the Safety and Immunogenicity of an Intranasal Vaccine for Respiratory Syncytial Virus in Seropositive Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meissa Vaccines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: MV-005
Record Dates: First submitted 2020-06-12; First posted 2020-06-23 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Live attenuated vaccine; Safety; Immunogenicity; Phase 1 clinical trial; Pediatric; Seropositive
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: The first 15 enrolled participants will be assigned to Dosage Group 1 and be randomly allocated to receive either investigational vaccine at Dosage 1 or placebo. The Safety Monitoring Committee will subsequently review Dosage Group 1 safety data through Day 14, to allow dosage escalation. The next 15 enrolled participants will be assigned to Dosage Group 2 and be randomly allocated to receive investigational vaccine at Dosage 2 or placebo. The Safety Monitoring Committee will subsequently review Dosage Group 2 safety data through Day 14, to allow dosage escalation. The final group (Dosage Group 3) will consist of up to 12 enrolled participants who will be allocated to receive investigational vaccine at Dosage 3.
Who Masked: Participant
Masking Description: The study is single-mask in 2 of the 3 dosage groups: study participants and their parent(s)/guardian(s) will not know their child's study assignment, whereas investigators, site staff, and site pharmacists will remain unmasked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dosage Group 1: RSV Vaccine Dosage 1 (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 1.
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 1)
- Dosage Group 1: Placebo (Placebo Comparator): Participants in this arm will receive a single intranasal dose of placebo.
  Interventions: Other: Placebo
- Dosage Group 2: RSV Vaccine Dosage 2 (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 2.
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 2)
- Dosage Group 2: Placebo (Placebo Comparator): Participants in this arm will receive a single intranasal dose of placebo.
  Interventions: Other: Placebo
- Dosage Group 3: RSV Vaccine Dosage 3 (Experimental): Participants in this arm will receive a single intranasal dose of the investigational RSV vaccine at Dosage 3.
  Interventions: Biological: Investigational RSV vaccine MV-012-968 (Dosage 3)

INTERVENTIONS:
Biological: Investigational RSV vaccine MV-012-968 (Dosage 1) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 1: RSV Vaccine Dosage 1
Biological: Investigational RSV vaccine MV-012-968 (Dosage 2) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 2: RSV Vaccine Dosage 2
Other: Placebo — Single dose administered intranasally on Day 1
  Arms: Dosage Group 1: Placebo; Dosage Group 2: Placebo
Biological: Investigational RSV vaccine MV-012-968 (Dosage 3) — Single dose administered intranasally on Day 1
  Arms: Dosage Group 3: RSV Vaccine Dosage 3

SUMMARY:
This study evaluates an investigational vaccine that is designed to protect humans against infection with respiratory syncytial virus (RSV) and is administered as drops in the nose. Specifically, the study analyzes the safety of, and the immune response to, the vaccine when administered to healthy children between the ages of 15 and 59 months who are seropositive to RSV.

ELIGIBILITY:
Key Inclusion Criteria:

1. Children aged 15-59 months
2. Good health based on history, physical examination and medical record review, without evidence or suspicion of chronic disease
3. Seropositive to RSV, as defined by serum neutralizing antibody titer above the threshold described in the study Analytical Plan
4. Written informed consent provided by parent(s)/guardian(s)

Key Exclusion Criteria:

1. Known or suspected chronic illness, particularly cardiopulmonary (including asthma or reactive airways disease), metabolic, hepatic, renal, or infectious (including recurrent or chronic sinusitis)
2. Known or suspected immunodeficiency
3. Household or close contact with anyone ≤ 6 months of age or with immunocompromised individual(s)
4. Nasal obstruction (including due to anatomic/structural causes, acute or chronic rhinosinusitis, or other causes)
5. Receipt of immunoglobulins, monoclonal antibodies and/or any blood products, or ribavirin within 3 months prior to study inoculation, or planned during study period
6. Receipt of an investigational RSV vaccine at any time
7. Any other condition that, in the judgment of the investigator, would be a risk to participant's safety and/or may interfere with study procedures or interpretation of results

Ages: 15 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2020-06-09 (Actual); Primary Completion 2021-05-07 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Solicited adverse events (AEs) | Immediate post-vaccination period
  Frequency of solicited AEs will be measured, categorized by severity. Solicited AEs are predefined AEs that may occur after investigational vaccine administration
Unsolicited AEs | Immediate post-vaccination period
  Frequency of unsolicited AEs will be measured, categorized by severity. Unsolicited AEs are any untoward medical occurrences in a participant administered the investigational vaccine, regardless of causal relationship to the investigational vaccine. Unsolicited AEs can include unfavorable and unintended signs (including abnormal laboratory findings), symptoms, or diseases temporally associated with the use of the investigational vaccine.
Serious adverse events (SAEs) | Full study duration, an average of 6 months
  Frequency of SAEs will be measured, categorized by vaccine-relatedness. SAEs are AEs, whether considered causally related to the investigational vaccine or not, that threaten life or result in any of the following: death, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or congenital anomaly/birth defect.
Medically attended adverse events (MAEs) | Full study duration, an average of 6 months
  Frequency of MAEs will be measured, categorized by vaccine-relatedness. MAEs are AEs, whether considered causally related to the investigational vaccine or not, with unscheduled medically attended visits, such as urgent care visits, acute primary care visits, emergency department visits, or other previously unplanned visits to a medical provider. Scheduled medical visits such as routine physicals, wellness checks, 'check-ups', and vaccinations, are not considered MAEs.

SECONDARY OUTCOMES:
Change in serum RSV-specific neutralizing antibody titers | Baseline through Day 28, an average of six (6) weeks
  Change in serum RSV-specific neutralizing antibody (nAb) titers will be measured per participant.
Change in serum binding (RSV F-specific) antibody titers | Baseline through Day 28, an average of six (6) weeks
  Change in serum binding (RSV F-specific) antibody titers will be measured per participant.
Change in nasal mucosal binding (RSV F-specific) antibody titers | Baseline through Day 28, an average of six (6) weeks
  Change in mucosal binding (RSV F-specific) antibody titers will be measured per participant.
Potential vaccine virus shedding: frequency | Baseline through Day 28, an average of four (4) weeks
  Frequency of any post-vaccination shedding of vaccine virus (as detected by viral culture) will be measured per dosage group and overall.
Potential vaccine virus shedding: magnitude | Baseline through Day 28, an average of four (4) weeks
  If post-vaccination shedding of vaccine virus is detected by culture, peak viral titer (measured in plaque forming units, PFU) will be measured per dosage group and overall.
Potential vaccine virus shedding: duration | Baseline through Day 28, an average of four (4) weeks
  If post-vaccination shedding of vaccine virus is detected by culture, duration of shedding (in days) will be measured per dosage group and overall.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Medzihradsky, MD MPH MS, Study Director — Meissa Vaccines, Inc.
Locations (3):
- United States (3):
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

REFERENCES:
- [Result] Stobart CC, Rostad CA, Ke Z, Dillard RS, Hampton CM, Strauss JD, Yi H, Hotard AL, Meng J, Pickles RJ, Sakamoto K, Lee S, Currier MG, Moin SM, Graham BS, Boukhvalova MS, Gilbert BE, Blanco JC, Piedra PA, Wright ER, Moore ML. A live RSV vaccine with engineered thermostability is immunogenic in cotton rats despite high attenuation. Nat Commun. 2016 Dec 21;7:13916. doi: 10.1038/ncomms13916. PMID 28000669